CLINICAL TRIAL: NCT03952845
Title: Tolerability of Intranasal Capsaicinoid Spray
Brief Title: Intranasal Capsaicinoid Spray
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1024481
Record Dates: First submitted 2019-05-11; First posted 2019-05-16 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Tolerance; Capsaicin; Rhinitis
Keywords: Capsaicin; Rhinitis
MeSH Terms: conditions — Rhinitis

STUDY DESIGN:
Intervention Model Description: In brief, three consecutive patients will receive the initial intervention dose, and complete a post-intervention assessment. Subsequent cohorts receive escalating doses that are determined in advance (see below). If no patients in the initial cohort experience a dose limiting toxicity, three new patients will be recruited into the subsequent cohort and each will receive the escalated dose. This process continues on until at least one patient in a cohort experiences a dose limiting toxicity. When this occurs, three new patients will be recruited but will receive the same dose as the patient who experienced a dose limiting toxicity. If no patients in this new cohort experience a dose limiting toxicity, three additional patients will be recruited and will receive the next predetermined escalated dose. However, if two of six patients experience a dose limiting toxicity, the trial is considered complete and the dose these six patients received is considered the maximum tolerated dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intranasal Capsaicin (Experimental): Separate patients will be given escalating doses of intranasal capsaicinoid spray
  Interventions: Other: Capsaicinoid

INTERVENTIONS:
Other: Capsaicinoid — This is a tolerability study on doses lower than previously published for the use of intranasal capsaicinoid in the treatment of rhinitis

SUMMARY:
Rhinitis is inflammation of the inside of the nose. Symptoms of rhinitis include itchiness, sneezing, and a "runny" nose (rhinorrhea). There are many different causes for rhinitis, including allergies, age, different irritants in the air, overacting nervous system, and others.

Many current treatments for rhinitis are not helpful or are unable to be used for long periods of time. Capsaicin ("Kap-Sey-Uh-Sin") is a natural product that is found in many spicy foods, including hot peppers. This natural product has been used as a lotion to prevent pain, and scientists have found that it may reduce the symptoms of rhinitis when used as a spray in the nose.

However, capsaicin is known to cause a burning sensation. This study is needed so we can figure out what doses of capsaicin cause this burning sensation, and to what level these doses cause discomfort. Capsaicin can also cause a small degree of tearing from the eyes when used as a spray in the nose, and can also cause the nose to become "runny" (rhinorrhea).

When the safest dose of capsaicin spray is found, that dose can be used to treat people with rhinitis that is not getting better from standard treatments.

DETAILED DESCRIPTION:
Inflammation of the nasal mucosa (internal lining of the nose) results in a condition called rhinitis. Patients with rhinitis suffer from nasal stuffiness, congestion, rhinorrhea (nasal discharge), sneezing, and itchiness. Rhinitis affects a large number of people, with several studies estimating that between 10 and 50% of people have rhinitis.

The term rhinitis includes many different diseases that are commonly divided into allergic rhinitis and non-allergic rhinitis. Allergic rhinitis is a result of allergen exposure, with the diagnosis requiring an identifiable offending agent. Common allergens include pollen, molds, animals, and insects. Allergic rhinitis has similar symptoms to those outlined above and can be confirmed by allergy skin testing. There is also a strong association between allergic rhinitis and asthma, with one third of allergic rhinitis patients also suffering from reactive airway disease.

On the other hand, non-allergic rhinitis is a broad category and includes all forms of rhinitis that do not have an identifiable allergic component. Subcategories of non-allergic rhinitis include occupational, gustatory, smoking, hormonal, senile, atrophic, medication-induced, vasomotor (idiopathic), local allergic, and non-allergic rhinitis with eosinophilia syndrome (NARES).

Avoidance of triggers and use of intranasal medication, such as intranasal steroids and intranasal antihistamines, are the mainstays of treatment for non-allergic rhinitis. Combination of intranasal steroid and antihistamine has recently been developed as a single product and approved for the use in both allergic and non-allergic rhinitis. When high volume, clear rhinorrhea is the primary rhinitis symptom, intranasal anticholinergics have shown good effect. Finally, surgical intervention is considered in patients with select non-allergic rhinitis causes, such as vasomotor rhinitis.

The use of intranasal capsaiscinoid spray for treatment of rhinitis has been investigated for many years. The first identifiable trial was in 1991 and showed that both subjective and objective measurements of chronic rhinitis were reduced with repeated applications of intranasal capsaicin.

Capsaicinoids are active ingredients in the plant genus Capsicum, which includes bell peppers, habanero peppers, and jalapeno peppers, amongst others. The most noteworthy of the capsaicinoids is capsaicin. All capsaicinoids are irritants for humans, and they give the Capsicum plants their pungent taste and hot sensation, as well as produce the burning sensation from topical application.

Capsaicinoids are believed to be effective for non-allergic rhinitis due to their ability to block specific nerve fibers in the lining of the nose. Blocking this pathway results in decreased nasal hypersensitivity and leads to reduced nasal obstruction, sneezing, and rhinorrhea.

More recently, a systematic review for the Cochrane Collaboration was carried out. Four studies were included in the review, representing 302 patients. The authors of the review conclude that given many therapeutic options for non-allergic rhinitis are ineffective, the use of intranasal capsaicinoid as possible treatment modality is reasonable.

It should be noted that each of the four studies included in the review utilized a different dose of capsaiscinoid, and indeed a different capsaiscinoid altogether.

Despite many trials documenting the efficacy of intranasal capsaicinoids for non-allergic rhinitis, tolerability of the intervention is poorly studied. Also of note is that many of the current studies utilizing intranasal capsaicinoids have used some form of topical anesthetic in order to deliver high doses.

Therefore, given that intranasal capsaicinoid spray is an enticing treatment option for non-allergic rhinitis in terms of efficacy, and there is a dearth of reliable tolerability studies, we would seek to identify the side effect profile of a naturally sourced intranasal capsaicin spray. As pelargonic acid vanillylamide (PAVA) is the most studied capsaicinoid in terms of efficacy in humans, we propose to utilize this for our study.

The proposed study would address the following objectives:

1. Determine the rate and severity of intranasal burning sensation and pain with administration of intranasal PAVA in an otherwise healthy population with no history of medical or surgical nasal disease

   a. Measured using both a Likert scale and a Visual Analogue Scale (VAS)
2. Determine the rate and severity of lacrimation with administration of intranasal PAVA in an otherwise healthy population with no history of medical or surgical nasal disease

   a. Measured using a Likert scale
3. Determine the rate and severity of rhinorrhea with administration of intranasal PAVA in an otherwise healthy population with no history of medical or surgical nasal disease

   a. Measured using a Likert scale
4. Determine the overall patient perceived tolerability of intranasal PAVA administration in an otherwise healthy population with no history of medical or surgical nasal disease a. Considered an overall combined measure of all Likert scales and VAS

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* American Association of Anesthesiology Class 1,"A normal, healthy patient" only

Exclusion Criteria:

* Age less than 18 years
* Pregnancy
* Previous nasal or paranasal sinus surgery or radiation
* Allergies to capsaicinoids or capsaicinoid containing products (any combination of sweet peppers, or hot peppers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2030-07-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain - Visual Analogue Scale (VAS) - Change from 1 hour after pre-treatment baseline | Pre-treatment and Immediate (1 hour after treatment)
  Visual analogue scale will be used to analyze participant's perception of pain with the use of intranasal capsaicinoid spray. The visual analogue scale will be presented as a single line scale that is 100mm (0mm to 100mm) in length that the patient my place a mark on to indicate the severity of their pain. The distance (mm) of this mark from the 0 set point will determine the severity score.
Pain - Visual Analogue Scale (VAS) - Change from 1 week after pre-treatment baseline | Pre-treatment and Delayed (1 week after treatment)
  Visual analogue scale will be used to analyze participant's perception of pain with the use of intranasal capsaicinoid spray. The visual analogue scale will be presented as a single line scale that is 100mm (0mm to 100mm) in length that the patient my place a mark on to indicate the severity of their pain. The distance (mm) of this mark from the 0 set point will determine the severity score.
Rhinorrhea - Likert - Change from 1 hour after pre-treatment baseline | Pre-treatment and Immediate (1 hour after treatment)
  Likert scale will be used to analyze participant's perception of rhinorrhea ("runny-nose") with the use of intranasal capsaicinoid spray. Likert scale choices include: None (0), Very minimal (1), Mild (2), Moderate (3), Severe (4), and Very severe (5). Only a single option may be chosen, and this will be used to determine the severity score.
Rhinorrhea - Likert - Change from 1week after pre-treatment baseline | Pre-treatment and Delayed (1 week after treatment)
  Likert scale will be used to analyze participant's perception of rhinorrhea ("runny-nose") with the use of intranasal capsaicinoid spray. Likert scale choices include: None (0), Very minimal (1), Mild (2), Moderate (3), Severe (4), and Very severe (5). Only a single option may be chosen, and this will be used to determine the severity score.
Lacrimation - Likert - Change from 1 hour after pre-treatment baseline | Pre-treatment and Immediate (1 hour after treatment)
  Likert scale will be used to analyze participant's perception of lacrimation ("teary-eyes") with the use of intranasal capsaicinoid spray. Likert scale choices include: None (0), Very minimal (1), Mild (2), Moderate (3), Severe (4), and Very severe (5). Only a single option may be chosen, and this will be used to determine the severity score.
Lacrimation - Likert - Change from 1 week after pre-treatment baseline | Pre-treatment and Delayed (1 week after treatment)
  Likert scale will be used to analyze participant's perception of lacrimation ("teary-eyes") with the use of intranasal capsaicinoid spray. Likert scale choices include: None (0), Very minimal (1), Mild (2), Moderate (3), Severe (4), and Very severe (5). Only a single option may be chosen, and this will be used to determine the severity score.
Pain - Likert - Change from 1 hour after pre-treatment baseline | Pre-treatment and Immediate (1 hour after treatment)
  Likert scale will be used to analyze participant's perception of pain with the use of intranasal capsaicinoid spray. Likert scale choices include: None (0), Very minimal (1), Mild (2), Moderate (3), Severe (4), and Very severe (5). Only a single option may be chosen, and this will be used to determine the severity score.
Pain - Likert - Change from 1 week after pre-treatment baseline | Pre-treatment and Delayed (1 week after treatment)
  Likert scale will be used to analyze participant's perception of pain with the use of intranasal capsaicinoid spray. Likert scale choices include: None (0), Very minimal (1), Mild (2), Moderate (3), Severe (4), and Very severe (5). Only a single option may be chosen, and this will be used to determine the severity score.

CONTACTS AND LOCATIONS:
Overall Officials: S Mark Taylor, MD FRCSC, Principal Investigator — Dalhousie University; David WA Forner, MD, Study Director — Dalhousie University
Locations (1):
- Queen Elizabeth II Health Science Center, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No